CLINICAL TRIAL: NCT01491893
Title: Dose-finding and Safety Study of an Oncolytic Polio/Rhinovirus Recombinant Against Recurrent WHO Grade IV Malignant Glioma
Brief Title: PVSRIPO for Recurrent Glioblastoma (GBM)
Acronym: PVSRIPO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Istari Oncology, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); Brain Tumor Research Charity Grant (Unknown); Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro00031169; NS20023 (Other Grant/Funding Number: National Institute of Neurological Disorders and Stroke)
Record Dates: First submitted 2011-12-01; First posted 2011-12-14 (Estimated); Results first posted 2018-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2022-06

CONDITIONS: GBM; Glioblastoma; Glioma; Malignant Glioma
Keywords: GBM; Brain Tumor; Poliovirus Vaccine; WHO Grade IV Malignant Glioma
MeSH Terms: conditions — Glioblastoma; Glioma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Dose Level 1 (dose escalation) (Experimental): Participants received a single intratumoral infusion of 1.0 x 10^8 TCID50 Recombinant nonpathogenic polio-rhinovirus chimera (PVSRIPO), via convection-enhanced delivery to the brain tumor, with 4 weeks of monitoring for toxicities after infusion.
  Interventions: Biological: Recombinant nonpathogenic polio-rhinovirus chimera (PVSRIPO)
- Dose Level 2 (dose escalation) (Experimental): Participants received a single intratumoral infusion of 3.3 x 10^8 TCID50 Recombinant nonpathogenic polio-rhinovirus chimera (PVSRIPO), via convention-enhanced delivery to the brain tumor, with 4 weeks of monitoring for toxicities after infusion.
  Interventions: Biological: Recombinant nonpathogenic polio-rhinovirus chimera (PVSRIPO)
- Dose Level 3 (dose escalation) (Experimental): Participants received a single intratumoral infusion of 1.0 x 10^9 TCID50 Recombinant nonpathogenic polio-rhinovirus chimera (PVSRIPO), via convection-enhanced delivery to the brain tumor, with 4 weeks of monitoring for toxicities after infusion.
  Interventions: Biological: Recombinant nonpathogenic polio-rhinovirus chimera (PVSRIPO)
- Dose Level 4 (dose escalation) (Experimental): Participants received a single intratumoral infusion of 3.3 x 10^9 TCID50 Recombinant nonpathogenic polio-rhinovirus chimera (PVSRIPO), via convection-enhanced delivery to the brain tumor, with 4 weeks of monitoring for toxicities after infusion.
  Interventions: Biological: Recombinant nonpathogenic polio-rhinovirus chimera (PVSRIPO)
- Dose Level 5 (dose escalation) (Experimental): Participants received a single intratumoral infusion of 1.0 x 10^10 TCID50 Recombinant nonpathogenic polio-rhinovirus chimera (PVSRIPO), via convection-enhanced delivery to the brain tumor, with 4 weeks of monitoring for toxicities after infusion.
  Interventions: Biological: Recombinant nonpathogenic polio-rhinovirus chimera (PVSRIPO)
- Dose Level 4 (dose de-escalation) (Experimental): Participants received a single intratumoral infusion of 3.3 x 10^9 TCID50 Recombinant nonpathogenic polio-rhinovirus chimera (PVSRIPO), via convection-enhanced delivery to the brain tumor, with 4 weeks of monitoring for toxicities after infusion.
  Interventions: Biological: Recombinant nonpathogenic polio-rhinovirus chimera (PVSRIPO)
- Dose Level 2 (dose expansion) (Experimental): Participants received a single intratumoral infusion of 3.3 x 10^8 TCID50 of PVSRIPO, via convection-enhanced delivery to the brain tumor, with 4 weeks of monitoring for toxicities after infusion.
  Interventions: Biological: Recombinant nonpathogenic polio-rhinovirus chimera (PVSRIPO)
- Dose Level -1 (dose expansion) (Experimental): Participants received a single intratumoral infusion of 5.0 x 10^7 TCID50 Recombinant nonpathogenic polio-rhinovirus chimera (PVSRIPO), via convection-enhanced delivery to the brain tumor, with 4 weeks of monitoring for toxicities after infusion.
  Interventions: Biological: Recombinant nonpathogenic polio-rhinovirus chimera (PVSRIPO)
- Dose Level -2 (dose expansion) (Experimental): Participants received a single intratumoral infusion of 1.0 x 10^7 TCID50 Recombinant nonpathogenic polio-rhinovirus chimera (PVSRIPO), via convection-enhanced delivery to the brain tumor, with 4 weeks of monitoring for toxicities after infusion.
  Interventions: Biological: Recombinant nonpathogenic polio-rhinovirus chimera (PVSRIPO)
- Dose Level -1 (selected dose expansion) (Experimental): Participants received a single intratumoral infusion of 5.0 x 10^7 TCID50 Recombinant nonpathogenic polio-rhinovirus chimera (PVSRIPO), via convection-enhanced delivery to the brain tumor, with 4 weeks of monitoring for toxicities after infusion.
  Interventions: Biological: Recombinant nonpathogenic polio-rhinovirus chimera (PVSRIPO)

INTERVENTIONS:
Biological: Recombinant nonpathogenic polio-rhinovirus chimera (PVSRIPO) — Recombinant nonpathogenic polio-rhinovirus chimera (PVSRIPO)
  Other Names: Live attenuated, oral (Sabin) serotype 1 poliovirus vaccine

SUMMARY:
Purpose of the Study:

To determine the maximally tolerated dose (MTD) and the Recommended Phase 2 Dose (RP2D) of PVSRIPO when delivered intracerebrally by convection-enhanced delivery (CED). To obtain correlative mechanistic evidence of PVSRIPO's effects on infected WHO Grade IV malignant glioma tumors and to estimate progression-free survival (PFS) and overall survival (OS) in recurrent WHO Grade IV malignant glioma patients. To obtain information about clinical response rates to intratumoral inoculation of PVSRIPO. To estimate the efficacy of PVSRIPO administered at the optimal dose.

DETAILED DESCRIPTION:
PVSRIPO is a genetically recombinant, non-pathogenic poliovirus:rhinovirus chimera with a tumor-specific conditional replication phenotype. It consists of the genome of the live attenuated poliovirus serotype 1 (SABIN) vaccine (PV1S) with its cognate internal ribosomal entry site (IRES) element replaced with that of human rhinovirus type 2 (HRV2). PVSRIPO has been manufactured at NCI-Frederick, NCI, NIH.

Catheter Implantation: PVSRIPO will be delivered directly into the tumor. A stereotactic biopsy will be performed prior to virus administration for frozen section confirmation of viable tumor and further analysis. The biopsy needle will be placed with stereotactic guidance by a Cosman-Robert-Wells, MRI-compatible, stereotactic head frame or similar frameless device. Immediately following the stereotactically-guided tumor biopsy, a catheter will be implanted in the operating room (OR) at a site the same or different from that used for the biopsy using sterile techniques. A CT may be used to confirm catheter placement post-operatively.

Agent infusion: The entire volume of the agent to be delivered will be pre-loaded into a syringe by the investigational pharmacist and connected to the catheter under sterile conditions in the Neuro-Surgical Intensive Care Unit (NSICU) or neuro step down unit just prior to the beginning of infusion. Drug infusion will occur in the NSICU or neuro step down unit so that all other emergency facilities will be available. Patients will be infused through a Medfusion 3500 or 3010 infusion pump pre-programmed to a delivery rate of 500 microliters/hour. The total amount of the inoculum delivered to the patient will be 3 ml. The virus injection procedure will be completed within 6.5 hours. The catheter will be removed following the post-PVSRIPO infusion MRI.

Biopsy sampling and analyses: Biopsy material will be obtained from tumor tissue prior to virus administration. This tissue material will be subjected to routine histology to confirm tumor recurrence by the study neuropathologist, Dr. R. McLendon or his designate. Molecular genetic tests will also be conducted on extracts of tumor cells from the protocol-specified biopsy prior to PVSRIPO infusion. After acquiring sufficient tissue for standard clinical pathologic testing, up to three additional core biopsies will be obtained, if possible. The additional core biopsies will be used for genetic analysis, including full genome or full exome sequencing, as well as other molecular genetic testing. This testing will include, but is not limited to, DNA sequencing, gene amplification, and gene expression. Additional pathology tests on the protocol-specified biopsy tissue may be included, if a sufficient amount of tissue remains after standard clinical pathologic testing.

Selected patients who benefited from the initial infusion of PVSRIPO within this protocol will be eligible for a second infusion. All procedures previously described will be followed; however, the addition of a single dose of lomustine 8 weeks after PVSRIPO administration will alter the schedule of events that was previously described.

During the dose escalation phase of the study, the starting amount (dose level 1) of PVSRIPO to be delivered was 1.0 x 10^8 tissue culture infectious dose (TCID50). Dose level 2 was 3.3 x 10^8 TCID50, dose level 3 was 1.0 x 10^9 TCID50, dose level 4 was 3.3 x 10^9 TCID50, and dose level 5 wase 1.0 x 10^10 TCID50. 50% Tissue Culture Infective Dose (TCID50) is the unit of measure of infectious virus titer.

To minimize the number of patients treated at low-dose levels during the dose escalation phase, we used a two-step continual reassessment method (CRM) design that included an escalation step and a model-guided step. In the dose escalation phase, dose levels were rapidly escalated as preclinical data suggested that dose-limiting toxicity (DLT) would not occur at any of the five dose levels that were being evaluated. Decisions concerning dose escalation for subsequent patients were based upon the occurrence of DLT during the first 4 weeks after treatment administration. Initially, each patient was observed for ≥ 4 weeks before the next patient was treated. Starting at dose level 1, one patient was to be treated at each higher dose level. If no DLT was observed within 4 weeks of administration, then the next patient was to be treated at the next higher dose. If no DLTs were observed among patients treated on the first four dose levels, subsequent patients were to be treated at dose level 5. The escalation step was to be interrupted if a patient assigned to one of the first 4 dose levels or more than 20% of patients treated at dose level 5 experienced a DLT. In that case, further dose escalation or de-escalation would be guided by the likelihood-based implementation of the CRM, in which the one-parameter hyperbolic tangent model would be used to estimate the probability of DLT at each of the 5 dose levels based upon available data. The highest dose level for which this estimated probability is less than 20% would be identified as the maximum tolerated dose (MTD).

After completion of the dose escalation phase and determination of the MTD, the study protocol was amended to allow continued patient accrual to a dose expansion phase, in order to aid in the determination of the Recommended Phase II Dose (RP2D), and to garner more information about patient safety. The RP2D of PVSRIPO is the safe, therapeutic dose where patients have not experienced undue side effects from PVSRIPO or from the management of cerebral inflammation secondary to PVSRIPO administration. To address difficulties tapering patients off of steriods, the dose was reduced to dose level 2 (3.3 x 10^8 TCID50) for the dose expansion phase. After 6 patients were treated at dose level 2 in the dose expansion phase, due to continued difficulties tapering patients off steroids, the protocol was amended to further reduce the dose to dose level -1 (5.0 x 10^7 TCID50) with the goal of limiting the occurrence of known possible side effects of prolonged steroid use in patients who otherwise benefit from this investigational therapy. After the treatment of 24 patients at dose level -1, despite the fact that these patients were able to remain off significant doses of steroids, the patients benefiting the most from PVSRIPO appeared to be those who had experienced minimal or easily controllable inflammation. Hence, the protocol was amended to reduce the PVSRIPO dose to dose level -2 (1.0 x 10^7 TCID50) with the goal of limiting the occurrence of undesirable burden from inflammation and its treatment on as many subjects (and caregivers) as possible. Based upon additional animal studies, dose level -2 (1.0 x 10^7 TCID50) would also be a therapeutic dose. Reduction to dose level -2 was not due to concerns for the safety of the patients on dose level -1, but due to the observation that less inflammatory reaction appeared to be a predictor of better survival and treatment response. After treating 15 patients at dose level -2, based upon pre-clinical and clinical data collected on dose levels -1 and -2, there was no evidence of pre-clinically or clinically important differences between these dose levels. Therefore, the decision was made to treat all future study patients at dose level -1 (5.0 x 10^7 TCID50).

ELIGIBILITY:
Inclusion Criteria:

1. Disease Status. Patients must have a recurrent supratentorial WHO Grade IV malignant glioma based on imaging studies with measurable disease (≥ 1 cm or ≤ 5.5 cm of contrast-enhancing tumor). Prior histopathology consistent with a World Health Organization (WHO) Grade IV malignant glioma confirmed by the study pathologist, Roger McLendon, or his designate.
2. Age. Due to the potential implications of the treatment on the developing CNS, all patients must be ≥ 18 years of age at the time of entry into the study.
3. Performance Status. The patient must have a Karnofsky Performance Score (KPS) of ≥ 70% at the time of entry.
4. Laboratory Studies

   * Platelet count ≥ 125,000/microliter prior to biopsy. Platelets ≥ 100,000/microliter prior to infusion
   * Prothrombin and Partial Thromboplastin Times ≤ 1.2 x normal prior to biopsy
   * Positive serum anti-poliovirus titer prior to biopsy (except for retreatment)
   * Creatinine ≤ 1.2 x normal prior to biopsy
   * Total bilirubin, SGOT, SGPT, alkaline phosphatase ≤ 2.5 x normal prior to biopsy
   * Neutrophil count ≥ 1000 prior to biopsy
   * Hemoglobin ≥ 9 prior to biopsy
5. Poliovirus Immunization Booster. The subject must have received a boost immunization with trivalent inactivated IPOL™ (Sanofi-Pasteur) at least 1 week prior to administration of the study agent.
6. Disease Confirmation. At the time of biopsy, prior to administration of virus, the presence of recurrent tumor must be confirmed by histopathological analysis.
7. Informed Consent. A signed informed consent form approved by the Duke University Institutional Review Board (IRB) will be required for patient enrollment into the study. Patients must be able to read and understand the informed consent document and must sign the informed consent indicating that they are aware of the investigational nature of this study.
8. Brain MRI. Able to undergo brain MRI with and without contrast

Exclusion Criteria:

1. Pregnancy. Because of the unknown risk of virus administration potentially affecting a developing fetus or growing infant, females who are pregnant or breast-feeding during the study period will be excluded. Adults of reproductive potential not employing an effective method of birth control will be excluded. Sexually active women of child bearing potential, whose partner is male, must use medically accepted birth control. Sexually active men, whose partner is a female of child bearing potential, must use a medically accepted birth control.
2. Disease Status. Because patients will receive drug intracerebrally, patients with an impending, life-threatening cerebral herniation syndrome, based on the assessment of the study neurosurgeons, Allan Friedman, John Sampson, or Peter Fecci, or their designate, will be excluded.
3. Medical Conditions. Because the potential toxicities from the agent being studied in this protocol may be similar to some known diseases or may be more dangerous in the context of certain known diseases, the following patients will be excluded to avoid confounding the study results:

   * Patients with an active infection requiring intravenous treatment or having an unexplained febrile illness (Tmax > 99.5 F/37.5 C).
   * Patients with known immunosuppressive disease or known human immunodeficiency virus infection.
   * Unstable or severe intercurrent medical conditions such as severe heart (New York Heart Association Class 3 or 4) or known lung (FEV1 < 50%) disease, uncontrolled diabetes mellitus.
   * Albumin allergy. Albumin is added to the agent as a stabilizer. Patients with a known allergy will be excluded.
   * Current or history of anaphylactic reaction to gadolinium. Gadolinium is used as contrast for the MRI.
4. Previous Poliomyelitis. A history of neurological complications due to poliovirus infection would imply previous virus replication in the CNS. Based on animal studies, previous exposure to poliovirus administered intracerebrally can reduce subsequent virus replication in the CNS.
5. Prior Therapy. Patients who have not recovered from the toxic effects of prior chemotherapy and/or radiation therapy will be excluded. Guidelines for this recovery period are dependent upon the specific therapeutic agent being used:

   * Patients may not have received chemotherapy or bevacizumab ≤ 4 weeks [except for nitrosourea (6 weeks) or metronomic dosed chemotherapy such as daily etoposide or cyclophosphamide (1 week)] prior to starting the study drug unless patients have recovered from side effects of such therapy.
   * Patients may not have received immunotherapy ≤ 4 weeks prior to starting the study drug unless patients have recovered from side effects of such therapy.
   * Patients may not be less than 12 weeks from radiation therapy, unless progressive d disease outside of the radiation field or 2 progressive scans at least 4 weeks apart or histopathologic confirmation
   * Patients must have completed all standard of care treatments including surgical procedure and radiation therapy (at least 59Gy):

     * If the MGMT promoter in their tumor is known to be unmethylated, patients are not mandated to have received chemotherapy prior to participating in this trial.
     * If the MGMT promoter in their tumor is known to be methylated or the MGMT promoter status is unknown at the time of screening, patients must have received at least one chemotherapy regimen prior to participating in this trial.
6. Location and Extent of Tumor. Because of the potential toxicities from the agent, patients with neoplastic lesions in the brainstem, cerebellum or spinal cord, radiological evidence of multifocal disease, or leptomeningeal disease. Patients with evidence of diffuse subependymal disease or tumor in the brainstem, cerebellum, spinal cord, or CSF will be excluded. Since the study agent is a local treatment, patients with radiological evidence of active (growing) multifocal disease, tumors extending into or crossing the corpus callosum or leptomeningeal disease, will be excluded.
7. Subjects must not have diagnosis of agammaglobulinemia. Patients with the following will be excluded:

   * Undetectable anti-tetanus toxoid IgG (except for retreatment)
   * Known history of agammaglobulinemia
8. Patient on greater than 4mg per day of dexamethasone within the 2 weeks prior to admission for PVSRIPO infusion
9. Patient has worsening steroid myopathy (history of gradual progression of bilateral proximal muscle weakness, and atrophy of proximal muscle groups)
10. Patients with prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin

Eligibility Criteria for Retreatment:

Subjects can be considered for PVSRIPO retreatment if they meet some of the pertinent inclusion and exclusion criteria above. In addition, the subject must also satisfy the following criteria:

* Patient must have benefited from initial treatment with PVSRIPO (i.e. be at least 12 months following their initial PVSRIPO infusion).
* Patient must have a recurrence of their supratentorial WHO grade IV malignant glioma based on imaging studies with measurable disease (≥ 1 cm of contrast-enhancing tumor).
* At the time of biopsy, prior to administration of virus, the presence of recurrent tumor must be confirmed by histopathological analysis, unless already proven within the last 3 months via tissue sampling (biopsy or resection).
* The patient must have received a new boost immunization with trivalent inactivated IPOL™ (Sanofi-Pasteur) at least 1 week and no more than 4 weeks prior to re-administration of the study agent. The boost immunization may be obtained locally, prior to signing consent, as long as the patient has been informed about this study procedure via phone script.
* A new signed informed consent form for retreatment approved by the Duke University Institutional Review Board (IRB) will be required for retreatment. Patients must be able to read and understand the informed consent document and must sign the informed consent indicating that they are aware of the investigational nature of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-04-25 (Actual); Primary Completion 2017-06-27 (Actual); Study Completion 2021-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Landi, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brown MC, Beasley GM, McKay ZP, Yang Y, Desjardins A, Randazzo DM, Landi D, Ashley DM, Bigner DD, Nair SK, Gromeier M. Intratumor childhood vaccine-specific CD4+ T-cell recall coordinates antitumor CD8+ T cells and eosinophils. J Immunother Cancer. 2023 Apr;11(4):e006463. doi: 10.1136/jitc-2022-006463. PMID 37072349
- [Derived] Desjardins A, Gromeier M, Herndon JE 2nd, Beaubier N, Bolognesi DP, Friedman AH, Friedman HS, McSherry F, Muscat AM, Nair S, Peters KB, Randazzo D, Sampson JH, Vlahovic G, Harrison WT, McLendon RE, Ashley D, Bigner DD. Recurrent Glioblastoma Treated with Recombinant Poliovirus. N Engl J Med. 2018 Jul 12;379(2):150-161. doi: 10.1056/NEJMoa1716435. Epub 2018 Jun 26. PMID 29943666
- See also: The Preston Robert Tisch Brain Tumor Center at Duke — https://tischbraintumorcenter.duke.edu/
- See also: Duke Cancer Institute Clinical Trials — http://www.dukecancerinstitute.org/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1 (Dose Escalation): Participants received a single intratumoral infusion of 1.0 x 10^8 TCID50 of PVSRIPO, via convection-enhanced delivery to the brain tumor, with 4 weeks of monitoring for toxicities after infusion.
- Dose Level 2 (Dose Escalation); Dose Level 2 (Dose Expansion): Participants received a single intratumoral infusion of 3.3 x 10^8 TCID50 of PVSRIPO, via convection-enhanced delivery to the brain tumor, with 4 weeks of monitoring for toxicities after infusion.
- Dose Level 3 (Dose Escalation): Participants received a single intratumoral infusion of 1.0 x 10^9 TCID50 of PVSRIPO, via convection-enhanced delivery to the brain tumor, with 4 weeks of monitoring for toxicities after infusion.
- Dose Level 4 (Dose Escalation); Dose Level 4 (Dose De-escalation): Participants received a single intratumoral infusion of 3.3 x 10^9 TCID50 of PVSRIPO, via convection-enhanced delivery to the brain tumor, with 4 weeks of monitoring for toxicities after infusion.
- Dose Level 5 (Dose Escalation): Participants received a single intratumoral infusion of 1.0 x 10^10 TCID50 of PVSRIPO, via convection-enhanced delivery to the brain tumor, with 4 weeks of monitoring for toxicities after infusion.
- Dose Level -1 (Dose Expansion); Dose Level -1 (Selected Dose Expansion): Participants received a single intratumoral infusion of 5.0 x 10^7 TCID50 of PVSRIPO, via convection-enhanced delivery to the brain tumor, with 4 weeks of monitoring for toxicities after infusion.
- Dose Level -2 (Dose Expansion): Participants received a single intratumoral infusion of 1.0 x 10^7 TCID50 of PVSRIPO, via convection-enhanced delivery to the brain tumor, with 4 weeks of monitoring for toxicities after infusion.
Period: Overall Study
Arm/Group | Dose Level 1 (Dose Escalation) | Dose Level 2 (Dose Escalation) | Dose Level 3 (Dose Escalation) | Dose Level 4 (Dose Escalation) | Dose Level 5 (Dose Escalation) | Dose Level 4 (Dose De-escalation) | Dose Level 2 (Dose Expansion) | Dose Level -1 (Dose Expansion) | Dose Level -2 (Dose Expansion) | Dose Level -1 (Selected Dose Expansion)
Started | 1 | 1 | 1 | 1 | 4 | 1 | 6 | 24 | 15 | 7
Completed | 1 | 1 | 1 | 1 | 4 | 1 | 6 | 24 | 15 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Recombinant Nonpathogenic Polio-Rhinovirus Chimera (PVSRIPO): All participants who received a dose of PVSRIPO at any dose level
Arm/Group | Recombinant Nonpathogenic Polio-Rhinovirus Chimera (PVSRIPO)
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 57
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 57
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 61

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD will be the highest dose level for which the probability that a dose escalation patient experiences a dose-limiting toxicity (DLT) is estimated to be less than 20%. Any Grade 3 or 4 toxicity that is not reversible within 2 weeks, or any life-threatening event, or treatment-related death will be considered a DLT. Any grade 2 or higher serious autoimmune toxicities particularly those affecting vital organs (e.g. cardiac, renal, CNS) will be considered a DLT. 50% Tissue Culture Infective Dose (TCID50) is the unit of measure of infectious virus titer.
  The MTD was determined based on the first 9 patients treated with PVSRIPO- 1 at dose level 1 (1.0 x 10e8 TCID50 (50% Tissue Culture Infectious Dose)), 1 at dose level 2 (3.3 x 10e8 TCID50), 1 at dose level 3 (1.0 x 10e9 TCID50), 2 at dose level 4 (3.3 x 10e9 TCID50), and 4 at dose level 5 (1.0 x 10e10 TCID50).
Time Frame: 28 days after administration of PVSRIPO
Population: All participants who received a dose of PVSRIPO at any dose level
Measure: Number; unit: 50% Tissue Culture Infectious Dose
Groups:
- Dose Escalation Patients: Dose Escalation Patients
Arm/Group | Dose Escalation Patients
Number analyzed (Participants) | 9
50% Tissue Culture Infectious Dose | 10,000,000,000

2. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: The number of dose escalation patients experiencing a dose-limiting toxicity (DLT) will be reported. Any grade 3 or any Grade 4 toxicity that is not reversible within 2 weeks, or any life-threatening event, or treatment-related death will be considered a DLT. Any grade 2 or higher serious autoimmune toxicities particularly those affecting vital organs (e.g. cardiac, renal, CNS) will also be considered a DLT.
Time Frame: 28 days after administration of PVSRIPO
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 (Dose Escalation) | Dose Level 2 (Dose Escalation) | Dose Level 3 (Dose Escalation) | Dose Level 4 (Dose Escalation) | Dose Level 5 (Dose Escalation)
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 4
Participants | 0 | 0 | 0 | 0 | 1

3. Primary Outcome: Recommended Phase 2 Dose (RP2D)
Description: The RP2D of PVSRIPO is the safe, therapeutic dose where patients have not experienced undue side effects from PVSRIPO or from the management of cerebral inflammation secondary to PVSRIPO administration. 50% Tissue Culture Infective Dose (TCID50) is the unit of measure of infectious virus titer.
Time Frame: 5 years
Measure: Number; unit: 50% Tissue Culture Infectious Dose
Groups:
- All Participants: All Participants
Arm/Group | All Participants
Number analyzed (Participants) | 61
50% Tissue Culture Infectious Dose | 50000000

ADVERSE EVENTS:
Time Frame: From PVSRIPO administration until a patient is taken off study for disease progression or the participant started a new treatment regimen (average of 10 months).
Description: This includes all adverse events regardless of attribution to study treatment from the time of PVSRIPO administration until the patient is taken off study or is retreated with PVSRIPO. For the reporting of adverse events per dose level, all patients receiving a specific dose were combined.
Groups:
- Dose Level 1 Patients: Participants received a single intratumoral infusion of 1.0 x 10^8 TCID50 of PVSRIPO, via convection-enhanced delivery to the brain tumor, with 4 weeks of monitoring for toxicities after infusion.
- Dose Level 2 Patients: Participants received a single intratumoral infusion of 3.3 x 10^8 TCID50 of PVSRIPO, via convection-enhanced delivery to the brain tumor, with 4 weeks of monitoring for toxicities after infusion.
- Dose Level 3 Patients: Participants received a single intratumoral infusion of 1.0 x 10^9 TCID50 of PVSRIPO, via convection-enhanced delivery to the brain tumor, with 4 weeks of monitoring for toxicities after infusion.
- Dose Level 4 Patients: Participants received a single intratumoral infusion of 3.3 x 10^9 TCID50 of PVSRIPO, via convection-enhanced delivery to the brain tumor, with 4 weeks of monitoring for toxicities after infusion.
- Dose Level 5 Patients: Participants received a single intratumoral infusion of 1.0 x 10^10 TCID50 of PVSRIPO, via convection-enhanced delivery to the brain tumor, with 4 weeks of monitoring for toxicities after infusion.
- Dose Level -1 Patients: Participants received a single intratumoral infusion of 5.0 x 10^7 TCID50 of PVSRIPO, via convection-enhanced delivery to the brain tumor, with 4 weeks of monitoring for toxicities after infusion.
- Dose Level -2 Patients: Participants received a single intratumoral infusion of 1.0 x 10^7 TCID50 of PVSRIPO, via convection-enhanced delivery to the brain tumor, with 4 weeks of monitoring for toxicities after infusion.
Arm/Group | Dose Level 1 Patients | Dose Level 2 Patients | Dose Level 3 Patients | Dose Level 4 Patients | Dose Level 5 Patients | Dose Level -1 Patients | Dose Level -2 Patients
All-Cause Mortality (participants affected / at risk) | 0/1 | 6/7 | 1/1 | 2/2 | 4/4 | 24/31 | 12/15
Serious Adverse Events (participants affected / at risk) | 1/1 | 3/7 | 1/1 | 1/2 | 3/4 | 7/31 | 5/15
Other Adverse Events (participants affected / at risk) | 1/1 | 7/7 | 1/1 | 2/2 | 4/4 | 31/31 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 Patients (N=1) | Dose Level 2 Patients (N=7) | Dose Level 3 Patients (N=1) | Dose Level 4 Patients (N=2) | Dose Level 5 Patients (N=4) | Dose Level -1 Patients (N=31) | Dose Level -2 Patients (N=15)
Cardiac arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Visual field cut - hemianopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatic hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Death NOS (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fever (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Steroid myopathy (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dystonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Edema cerebral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 1
Pyramidal tract syndrome (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 2 | 3
Seizure (Nervous system disorders) | 1 | 2 | 1 | 0 | 1 | 4 | 2
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 2
Delusions (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 3 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 Patients (N=1) | Dose Level 2 Patients (N=7) | Dose Level 3 Patients (N=1) | Dose Level 4 Patients (N=2) | Dose Level 5 Patients (N=4) | Dose Level -1 Patients (N=31) | Dose Level -2 Patients (N=15)
Anemia (Blood and lymphatic system disorders) | 1 | 4 | 1 | 2 | 3 | 19 | 11
Cardiac arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear and labyrinth disorders (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Cushingoid (Endocrine disorders) | 0 | 2 | 0 | 1 | 1 | 1 | 0
Diabetes (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blurred vision (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 3 | 1
Diplopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0
Eye disorders - Other, specify (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Farsighted (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Focusing difficulty (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Strabismus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Visual field cut - hemianopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 9 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 7 | 4
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 8 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 3 | 0 | 1 | 0 | 13 | 3
Taste disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 0 | 6 | 2
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Edema face (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 3 | 1 | 2 | 2 | 11 | 3
Fever (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 1 | 0 | 0 | 4 | 1
Infusion related reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Irritability (General disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 3 | 0 | 0 | 0 | 14 | 5
Steroid myopathy (General disorders) | 0 | 2 | 1 | 2 | 0 | 2 | 1
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Bronchial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis infective (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 2 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 3
Phlebitis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 9 | 6
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 3 | 2
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 1 | 1
Burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 4 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 1 | 0 | 5 | 4
Alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 3 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 0 | 2 | 0 | 9 | 4
Blood bilirubin increased (Investigations) | 0 | 2 | 0 | 1 | 0 | 1 | 2
Creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 7 | 2
Lymphocyte count decreased (Investigations) | 0 | 1 | 1 | 1 | 2 | 13 | 7
Neutrophil count decreased (Investigations) | 0 | 2 | 0 | 0 | 1 | 5 | 3
Platelet count decreased (Investigations) | 0 | 4 | 1 | 2 | 1 | 9 | 6
White blood cell decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 7 | 3
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 6 | 1 | 1 | 2 | 22 | 5
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 4 | 1 | 1 | 3 | 18 | 8
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 4 | 1 | 1 | 2 | 13 | 7
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 7 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 2 | 1 | 9 | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 3 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 2 | 10 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 5 | 1 | 0 | 0 | 7 | 3
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphasia (Nervous system disorders) | 0 | 2 | 1 | 0 | 2 | 13 | 2
Dystonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Facial muscle weakness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 5 | 0 | 2 | 1 | 23 | 9
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Myokymia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1
Paresthesia (Nervous system disorders) | 0 | 3 | 0 | 1 | 1 | 8 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyramidal tract syndrome (Nervous system disorders) | 0 | 2 | 0 | 1 | 3 | 18 | 8
Restless leg syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 6 | 1 | 0 | 3 | 15 | 10
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 5 | 0
Confusion (Psychiatric disorders) | 0 | 2 | 0 | 0 | 1 | 7 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 1
Hallucinations (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 4 | 0 | 0 | 1 | 8 | 2
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 5 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal calculi (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 4 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Irregular menstruation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 4 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 3 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 5 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 8 | 3
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin trauma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 2
Menopause (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hot flashes (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 8 | 3
Thromboembolic event (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-25): https://cdn.clinicaltrials.gov/large-docs/93/NCT01491893/Prot_SAP_000.pdf